CLINICAL TRIAL: NCT05666531
Title: Research on Innovative Diagnosis and Treatment System of Syndrome Differentiation of Zang-fu Viscera and Effectiveness Evaluation Based on Inter-Arm Blood Pressure Measured Simultaneously
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liyun He (Other)
Collaborators: Beijing University of Chinese Medicine (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Affiliated Hospital of Inner Mongolia Minzu University (Unknown); Hohhot Hospital of Mongolian Medicine and TCM (Unknown)
Responsible Party: Sponsor-Investigator, Liyun He, Director of TCM Clinical Efficacy Evaluation Center, China Academy of Chinese Medical Sciences
Organization: China Academy of Chinese Medical Sciences (Other)
Other Study IDs: 2022-1-4301
Record Dates: First submitted 2022-12-10; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Insomnia; Chronic Gastritis
Keywords: Blood pressure in both arms; syndrome differentiation; liver-spleen disharmony; efficacy evaluation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy people: The physical examination ruled out the disease
- Chronic gastritis: The endoscopic diagnosis is consistent with chronic gastritis or self-reported stomachache
- Insomnia: The Pittsburgh Sleep Quality Index Scale was measured and assessed as meeting a diagnosis of insomnia disorder or self-reported insomnia for more than three months

SUMMARY:
By combining the measurement of blood pressure in both arms with the information of the four diagnoses of TCM, we try to form a diagnostic model of "five diagnoses combined with ginseng" based on TCM Zang-fu syndrome differentiation. It can further objectify and visualize the fuzzy four diagnostic indicators of TCM. In order to solve the problem of data differentiation of TCM four diagnoses, and optimize the five diagnoses of TCM conjunctive index, explore the establishment of TCM intelligent diagnosis and treatment and contact evaluation computer system

ELIGIBILITY:
Inclusion Criteria:

Case inclusion Criteria:

* Patients were treated with epigastric pain and / or insomnia, which met the above diagnostic criteria for diseases, liver and spleen;
* diagnostic criteria for diseases, liver and spleen;
* Age 18-65 years old;
* It can combine mild and moderate depression, anxiety Sign the informed consent form.

Healthy control inclusion criteria:

* PSQI < 5 points;
* No hypertension, diabetes, hyperlipidemia, coronary heart disease and other underlying diseases;
* No depression, anxiety, malignant tumor, syphilis, HIV and other infectious diseases;
* Over 18 years of age;
* Volunteer to participate in this study, cooperate with the measurement of blood pressure in both arms, and sign the informed consent.

Exclusion Criteria:

Case exclusion criteria:

* Patients with insomnia disorder caused by uneffectively controlled or serious diseases, such as malignant tumor, persistent pain, cardiovascular and cerebrovascular diseases, endocrine diseases, etc.;
* patients with severe depression and mental illness;
* Pregnant and lactation patients.

Healthy controls exclusion criteria:

* sleep apnea syndrome or restless leg syndrome and other sleep disorders;
* Pregnant and lactation;
* Abnormal symptoms and abnormal tongue pulse occur in the body, such as facial acne, dysmenorrhea, thick and greasy tongue coating, loose stools, fat tongue, teeth marks and tongue.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical examination center and Hospital Outpatient Clinic
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure measurement in both arms | 5minutes
  The systolic blood pressure, diastolic blood pressure and pulse rate of the left and right upper arms were simultaneously measured by a standard dual-arm electronic sphygmomanometer. A total of 6 data were collected. A total of 30 data were collected and measured for 5 times without interruption, which was used to judge the functional balance state of "Zang-fu regional tissues" in human body.

SECONDARY OUTCOMES:
Pulse diagnosis information | 10minutes
  The data collected by tongue pulse analyzer were used as one of the diagnostic information of hepatic and splenic dysregulation
Pittsburgh Sleep Quality Index (PSQI） | 5minutes
  Pittsburgh Sleep Quality Index (PSQI）,used to assess the actual sleep status in the last 1 month.The total score ranges from 0 to 2l, with higher scores indicating poorer sleep quality
Hamilton Anxiety Scale (HAMA) | 5minutes
  Hamilton Anxiety Scale (HAMA),used to assess the severity of anxiety symptoms.The total score ranges from 0 to 56, with higher scores indicating more anxiety.
Hamilton Depression Scale (HAMD) | 5minutes
  Hamilton Depression Scale (HAMD), used to assess the severity of depression.The total score ranges from 0 to 96, with higher scores indicating more severe depression.
Gastrointestinal Symptom Scale | 5minutes
  Gastrointestinal Symptom Rating Scale (GSRS),used to assess gastrointestinal function for nearly one week.The total score ranges from 0 to 112, with higher scores indicating more severe gastrointestinal symptoms.
Grade table of main disorders of liver and spleen | 5minutes
  Grade table of main disorders of liver and spleen, used to assess the severity of the disorder of liver and spleen. The total score ranges from 0 to 24, with higher scores indicating more severe disorder of liver and spleen.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Shijitan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No